CLINICAL TRIAL: NCT05044195
Title: A Phase 3, Randomized, Observer-blind, Controlled, Multicenter, Clinical Study to Evaluate Immunogenicity and Safety of an MF59-adjuvanted Quadrivalent Subunit Inactivated Influenza Vaccine in Comparison With a Licensed Quadrivalent Influenza Vaccine, in Adults 50 to 64 Years of Age
Brief Title: A Clinical Study to Evaluate the Immunogenicity and Safety of an Adjuvanted Quadrivalent Influenza Vaccine Compared With a Licensed Quadrivalent Vaccine in Adults 50 to 64 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V118_23
Record Dates: First submitted 2021-09-06; First posted 2021-09-14 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-05

CONDITIONS: Influenza, Human
Keywords: Influenza, Vaccine, MF59 adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- aQIV (Experimental): Adjuvanted QIV containing 2 influenza type A strains and 2 influenza type B strains
  Interventions: Biological: aQIV
- Comparator QIV (Active Comparator): Non-adjuvanted comparator QIV containing 2 influenza type A strains and 2 influenza type B strains
  Interventions: Biological: Comparator QIV

INTERVENTIONS:
Biological: aQIV — Participants receive a 0.5-mL intramuscular dose of aQIV on Day 1
  Arms: aQIV
Biological: Comparator QIV — Participants receive a 0.5-mL intramuscular dose of Comparator QIV on Day 1
  Arms: Comparator QIV

SUMMARY:
This Phase 3 study is a randomized, observer-blind immunogenicity and safety study of aQIV (an MF59-adjuvanted quadrivalent influenza vaccine) compared with a licensed quadrivalent influenza vaccine in adults 50 to 64 years of age.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, all subjects must meet ALL of the following inclusion criteria:

* Individuals 50 to 64 years of age (i.e. 50 to ≤64 years) on the day of informed consent
* Individuals who have voluntarily given written consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry
* Individuals who can comply with study procedures including follow-up
* Males, females of non-childbearing potential or females of childbearing potential who are using an effective birth control method, at least 30 days prior to informed consent, which they intend to use for at least 2 months after the study vaccination

Exclusion Criteria:

In order to participate in this study, all subjects must not meet ANY of the exclusion criteria described below:

* Females of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of contraceptive methods from at least 30 days prior to study entry and who do not plan to do so until 2 months after the study vaccination
* Progressive, unstable or uncontrolled clinical conditions
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study
* History of any medical condition considered an AESI
* Known history of Guillain Barré syndrome or another demyelinating disease such as encephalomyelitis and transverse myelitis
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws
* Abnormal function of the immune system resulting from:

  1. Clinical conditions
  2. Systemic administration of corticosteroids (PO/IV/IM) at a dose equivalent to ≥20 mg/day of prednisone for more than 14 consecutive days within 90 days prior to informed consent. Topical, inhaled and intranasal corticosteroids are permitted. Intermittent use (one dose in 30 days) of intra-articular corticosteroids is also permitted
  3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent
* Received immunoglobulins or any blood products within 180 days prior to informed consent
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent, or who are unwilling to refuse participation in another clinical study at any time during the conduct of this study (notes: i. concomitant participation in a study not involving or no longer involving administration of drugs, vaccines, or medical devices, is acceptable (e.g. studies in safety follow-up phase, observational studies); ii. concomitant participation in a COVID-19 vaccine study is acceptable provided that the vaccine dosing interval mentioned in Exclusion Criterion #11 is adhered to)
* Receipt of any influenza vaccine within 6 months prior to enrollment in this study, or plan to receive influenza vaccine during the study period
* Receipt of any (investigational or licensed) COVID-19 vaccine within 14 days (non-replicating vaccines) or 28 days (replicating vaccines) prior to enrollment or plan to receive any COVID-19 vaccine within 7 days from study vaccination
* Receipt of any inactivated non-influenza vaccine within 14 days or live-attenuated vaccine within 28 days prior to enrollment in this study or plan to receive any other non-influenza vaccine within 28 days from study vaccination
* Acute (severe) febrile illness
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study
* Study personnel or immediate family members or household member of study personnel

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2044 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (29):
- United States (12):
  - 84013 Coastal Clinical Research, Inc., Mobile, Alabama
  - 84007 Alliance for Multispecialty Research, Tempe, Arizona
  - 84005 JEM Research Institute, Atlantis, Florida
  - 84010 Headlands Research Orlando, Orlando, Florida
  - 84001 Meridian Clinical Research, Savannah, Georgia
  - 84003 Meridian Clinical Research, Sioux City, Iowa
  - 84006 Alliance for Multispecialty Research, Kansas City, Missouri
  - 84009 Meridian Clinical Research, Lincoln, Nebraska
  - 84002 Meridian Clinical Research, Norfolk, Nebraska
  - 84004 Meridian Clinical Research, Omaha, Nebraska
  - 84008 United Medical Associates, Binghamton, New York
  - 84011 Meridian Clinical Research, Endwell, New York
- Estonia (6):
  - 23302 Vee Family Doctors Centre, Paide
  - 23301 Innomedica OÜ - Outpatient, Tallinn
  - 23303 Al Mare Perearstikeskus OÜ, Tallinn
  - 23304 Merelahe Family Doctors Centre, Tallinn
  - 23306 Center for Clinical and Basic Research, Tallinn
  - 23305 Clinical Research Center - Vaccine Trials, Tartu
- Germany (11):
  - 27602 Klinische Forschung Berlin, Berlin
  - 27603 Emovis GmbH, Berlin
  - 27608 Klinische Forschung Dresden GmbH, Dresden
  - 27609 IKF Pneumologie GmbH & Co. KG, Frankfurt
  - 27611 Siteworks GmbH, Fulda
  - 27601 Klinische Forschung Hamburg GmbH, Hamburg
  - 27605 Clinical Research Hamburg GmbH, Hamburg
  - 27604 Klinische Forschung Hannover-Mitte GmbH, Hanover
  - 27607 Siteworks GmbH, Hanover
  - 27606 SIBAmed GmbH & Co KG, Leipzig
  - 27610 Studienzentrum Leitz Triderm, Stuttgart

IPD SHARING:
Plan to Share IPD: Yes
SEQIRUS supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the CTD modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., ICH E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR])).
Supporting Information: Study Protocol, SAP
Time Frame: SEQIRUS discloses results from clinical studies within 12 months of last patient last visit (LPLV) unless otherwise mandated by local laws or regulations.
Access Criteria: SEQIRUS will consider requests from qualified scientific and medical researchers to disclose protocols, anonymized subject-level data and study-level data when there is medical, scientific and/or public health interest to ensure the safe use of a Seqirus product licensed on or after 1 January 2014 in the United States (US) and/or the European Union (EU). This applies to Seqirus-sponsored interventional studies initiated after 27 September 2007 and ongoing as of 26 December 2007, that have been included as part of a US or EU submission package which received approval in US and EU on or after 1 January 2014 and have been accepted for publication.
URL: https://www.seqirus.us/partnering

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the 2021/2022 Northern Hemisphere influenza season from 29 centers in Estonia (6 centers), Germany (11 centers), and the United States (12 centers).
Pre-assignment Details: In total, 2044 subjects were enrolled in the study.
Period: Overall Study
Arm/Group | aQIV | Comparator QIV
Started | 1027 | 1017
Received Study Vaccine | 1027 | 1016
Completed | 982 | 989
Not Completed | 45 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aQIV | Comparator QIV | Total
Number analyzed (Participants) | 1027 | 1017 | 2044
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1027 | 1017 | 2044
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (4.17) | 57.8 (4.21) | 57.8 (4.19)
Age, Customized [Count of Participants; unit: Participants]
  50 to 59 years | 609 | 596 | 1205
  60 to 64 years | 418 | 421 | 839
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 635 | 615 | 1250
  Male | 392 | 402 | 794
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 26
  Not Hispanic or Latino | 1013 | 1001 | 2014
  Unknown or Not Reported | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 2 | 4 | 6
  Black or African American | 39 | 36 | 75
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 982 | 972 | 1954
  Other | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 377 | 367 | 744
  Germany | 259 | 254 | 513
  Estonia | 391 | 396 | 787
Received an influenza vaccination in the previous 3 influenza seasons [Count of Participants; unit: Participants]
  Yes | 586 | 598 | 1184
  No | 441 | 419 | 860
Comorbidity Risk Score [Count of Participants; unit: Participants] — A subject's comorbidity risk score was obtained by adding scores for each applicable characteristic: age (<70; 70-74; 75-79; 80-89; ≥90 years); sex (female; male); number of outpatient visits during the previous year (0; 1-6; 7-12; ≥13); previous hospitalization due to pneumonia or influenza (no; yes); pre-existing comorbidity (pulmonary disease; heart disease; renal disease or renal transplant; dementia or stroke; nonhematological and hematological cancer). A cut-off score ≥50 defines higher probability of hospitalization due to pneumonia/influenza or death (Hak et al, J Infect Dis 2004).
  Participants
    <50 | 912 | 919 | 1831
    ≥50 | 115 | 98 | 213

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) and GMT Ratio of Hemagglutination Inhibition (HI) Antibodies at Day 22 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: The GMT ratio is defined as the geometric mean of the postvaccination HI titer for Comparator QIV over the geometric mean of the postvaccination HI titer for aQIV.
Time Frame: Day 22
Population: Per Protocol Set (PPS) Immunogenicity, defined as all subjects in the Full Analysis Set (FAS) Immunogenicity who: had both Day 1 and Day 22 immunogenicity assessment; correctly received the vaccine (ie, received the vaccine to which the subjects were randomized and at the scheduled time points); had no protocol deviations leading to exclusion as defined prior to unblinding/analysis; were not excluded due to other reasons defined prior to unblinding or analysis. Note: Adjusted GMTs are presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 983 | 985
Titer
  A/H1N1 | 731.90 [689.39 to 777.04] | 586.85 [552.83 to 622.96]
  A/H3N2 | 347.89 [324.78 to 372.64] | 313.16 [292.42 to 335.36]
  B/Yamagata | 154.40 [146.80 to 162.40] | 145.74 [138.57 to 153.27]
  B/Victoria | 144.41 [136.97 to 152.26] | 143.32 [135.97 to 151.07]
Statistical Analysis 1: Comparison: aQIV vs Comparator QIV; A/H1N1; Test type: Non-Inferiority — Non-inferiority criteria for the GMT ratio: upper limit (UL) of the 95% confidence interval (CI) for the inter-group GMT ratio is ≤1.5 for each vaccine strain; GMT ratio = 0.802, 95% CI 2-sided [0.738 to 0.871]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; A/H3N2; Test type: Non-Inferiority — Non-inferiority criteria for the GMT ratio: UL of the 95% CI for the inter-group GMT ratio is ≤1.5 for each vaccine strain; GMT ratio = 0.900, 95% CI 2-sided [0.819 to 0.989]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; B/Yamagata; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 0.944, 95% CI 2-sided [0.880 to 1.012]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; B/Victoria; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 0.992, 95% CI 2-sided [0.923 to 1.067]

2. Primary Outcome: Immunogenicity Endpoint: Seroconversion Rate (SCR) and SCR Difference for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: The SCR defined as the percentage of subjects with either a prevaccination HI titer <1:10 and a postvaccination (Day 22) HI titer ≥1:40, or with either a prevaccination HI titer ≥1:10 and a ≥4-fold increase in postvaccination HI titer.
  The SCR difference is defined as the Comparator QIV SCR minus the aQIV SCR.
Time Frame: Day 1 to Day 22
Population: PPS Immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 983 | 985
percentage of participants
  A/H1N1 | 81.2 [78.57 to 83.58] | 76.8 [74.04 to 79.42]
  A/H3N2 | 63.6 [60.46 to 66.63] | 61.8 [58.61 to 64.82]
  B/Yamagata | 43.4 [40.27 to 46.60] | 41.0 [37.92 to 44.19]
  B/Victoria | 44.5 [41.39 to 47.74] | 40.6 [37.52 to 43.76]
Statistical Analysis 1: Comparison: aQIV vs Comparator QIV; A/H1N1; Test type: Non-Inferiority — Non-inferiority criteria for the SCR difference: UL of the 95% CI for the difference in SCR is ≤10% for each vaccine strain; SCR difference = -4.4, 95% CI 2-sided [-7.97 to -0.74]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; A/H3N2; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference = -1.8, 95% CI 2-sided [-6.14 to 2.48]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; B/Yamagata; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference = -2.4, 95% CI 2-sided [-6.77 to 2.00]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; B/Victoria; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; SCR difference = -3.9, 95% CI 2-sided [-8.31 to 0.45]

3. Primary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio of HI Antibodies at Day 22 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: as for outcome 1
Time Frame: Day 22
Population: FAS Immunogenicity, defined as all subjects in the All Enrolled Set who were randomized, received study vaccination and provided immunogenicity data at any time point. Note: Adjusted GMTs are presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Titer
  A/H1N1 | 729.17 [687.51 to 773.36] | 589.07 [555.25 to 624.94]
  A/H3N2 | 347.09 [324.44 to 371.33] | 315.69 [295.04 to 337.79]
  B/Yamagata | 155.19 [147.67 to 163.09] | 146.89 [139.74 to 154.40]
  B/Victoria | 143.73 [136.44 to 151.42] | 143.74 [136.42 to 151.45]
Statistical Analysis 1: Comparison: aQIV vs Comparator QIV; A/H1N1; Test type: Superiority; GMT ratio = 0.808, 95% CI 2-sided [0.745 to 0.876]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; A/H3N2; Test type: Superiority; GMT ratio = 0.910, 95% CI 2-sided [0.829 to 0.998]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; B/Yamagata; Test type: Superiority; GMT ratio = 0.947, 95% CI 2-sided [0.884 to 1.014]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; B/Victoria; Test type: Superiority; GMT ratio = 1.000, 95% CI 2-sided [0.931 to 1.075]

4. Secondary Outcome: Immunogenicity Endpoint: GMT and GMT Ratio of HI Antibodies at Day 181 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: as for outcome 1
Time Frame: Day 181
Population: FAS Immunogenicity. Note: Adjusted GMTs are presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Titer
  A/H1N1 | 351.73 [331.61 to 373.06] | 306.11 [288.62 to 324.66]
  A/H3N2 | 165.17 [155.85 to 175.05] | 157.34 [148.48 to 166.73]
  B/Yamagata | 83.42 [79.81 to 87.20] | 84.53 [80.87 to 88.36]
  B/Victoria | 79.51 [75.81 to 83.40] | 81.73 [77.92 to 85.72]
Statistical Analysis 1: Comparison: aQIV vs Comparator QIV; A/H1N1; Test type: Other; GMT ratio = 0.870, 95% CI 2-sided [0.803 to 0.944]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; A/H3N2; Test type: Other; GMT ratio = 0.953, 95% CI 2-sided [0.880 to 1.032]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; B/Yamagata; Test type: Other; GMT ratio = 1.013, 95% CI 2-sided [0.953 to 1.077]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; B/Victoria; Test type: Other; GMT ratio = 1.028, 95% CI 2-sided [0.963 to 1.098]

5. Secondary Outcome: Immunogenicity Endpoint: GMT of HI Antibodies on Day 1, Day 22, and Day 181 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: GMTs on Day 1 (prior to vaccination), Day 22 (3 weeks after vaccination), and Day 181 (6 months after vaccination) as determined by HI assay against each of the four vaccine strains
Time Frame: Day 1 to Day 181
Population: FAS Immunogenicity. Note: Unadjusted GMTs are presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Titer
  A/H1N1 Day 1 GMT | 54.37 [49.71 to 59.47] | 50.41 [46.13 to 55.09]
  A/H1N1 Day 22 GMT | 708.36 [666.39 to 752.98] | 553.70 [519.14 to 590.56]
  A/H1N1 Day 181 GMT | 330.76 [308.44 to 354.70] | 276.24 [257.32 to 296.56]
  A/H3N2 Day 1 GMT | 45.97 [42.06 to 50.25] | 46.54 [42.63 to 50.81]
  A/H3N2 Day 22 GMT | 323.40 [300.77 to 347.73] | 292.50 [271.72 to 314.88]
  A/H3N2 Day 181 GMT | 151.92 [141.27 to 163.37] | 143.80 [133.33 to 155.09]
  B/Yamagata Day 1 GMT | 38.50 [35.83 to 41.38] | 38.33 [35.68 to 41.18]
  B/Yamagata Day 22 GMT | 144.30 [136.02 to 153.08] | 134.15 [126.31 to 142.48]
  B/Yamagata Day 181 GMT | 76.87 [72.33 to 81.70] | 77.34 [72.72 to 82.25]
  B/Victoria Day 1 GMT | 36.24 [33.78 to 38.87] | 37.06 [34.56 to 39.73]
  B/Victoria Day 22 GMT | 134.45 [126.24 to 143.21] | 132.45 [124.32 to 141.10]
  B/Victoria Day 181 GMT | 74.17 [69.66 to 78.97] | 75.99 [71.42 to 80.85]

6. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Fold Increase (GMFI) for Day 22/Day 1 and Day 181/Day 1 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: The GMFI is defined as the geometric mean of the fold increase of postvaccination HI titer over the prevaccination HI titer.
Time Frame: Day 1 to Day 181
Population: FAS Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Fold Increase
  A/H1N1 Fold increase Day 22 HI Titer | 13.07 [11.92 to 14.34] | 11.00 [10.07 to 12.02]
  A/H1N1 Fold increase Day 181 HI Titer | 6.22 [5.71 to 6.76] | 5.47 [5.03 to 5.95]
  A/H3N2 Fold increase Day 22 HI Titer | 7.09 [6.43 to 7.83] | 6.31 [5.78 to 6.89]
  A/H3N2 Fold increase Day 181 HI Titer | 3.29 [3.04 to 3.56] | 3.08 [2.86 to 3.31]
  B/Yamagata Fold increase Day 22 HI Titer | 3.77 [3.50 to 4.07] | 3.50 [3.25 to 3.77]
  B/Yamagata Fold increase Day 181 HI Titer | 2.03 [1.91 to 2.16] | 2.01 [1.89 to 2.14]
  B/Victoria Fold increase Day 22 HI Titer | 3.73 [3.45 to 4.02] | 3.60 [3.33 to 3.88]
  B/Victoria Fold increase Day 181 HI Titer | 2.06 [1.93 to 2.19] | 2.05 [1.92 to 2.20]

7. Secondary Outcome: Immunogenicity Endpoint: The Percentage of Subjects With a Titer ≥1:40 at Day 1, Day 22, and Day 181 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: Percentage of subjects with a titer ≥1:40 on Day 1, Day 22, and Day 181 as determined by HI assay against each of the four vaccine strains
Time Frame: Day 1 to Day 181
Population: FAS Immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
percentage of participants
  A/H1N1 HI Titer ≥1:40 at Day 1 | 65.2 [62.20 to 68.15] | 64.2 [61.14 to 67.15]
  A/H1N1 HI Titer ≥1:40 at Day 22 | 99.7 [99.14 to 99.94] | 99.2 [98.44 to 99.66]
  A/H1N1 HI Titer ≥1:40 at Day 181 | 98.2 [97.13 to 98.92] | 96.3 [94.89 to 97.36]
  A/H3N2 HI Titer ≥1:40 at Day 1 | 60.3 [57.16 to 63.30] | 61.7 [58.61 to 64.72]
  A/H3N2 HI Titer ≥1:40 at Day 22 | 97.5 [96.39 to 98.40] | 97.3 [96.12 to 98.23]
  A/H3N2 HI Titer ≥1:40 at Day 181 | 92.0 [90.08 to 93.59] | 89.9 [87.81 to 91.68]
  B/Yamagata HI Titer ≥1:40 at Day 1 | 60.8 [57.77 to 63.87] | 61.9 [58.81 to 64.90]
  B/Yamagata HI Titer ≥1:40 at Day 22 | 95.9 [94.47 to 97.01] | 94.6 [93.05 to 95.94]
  B/Yamagata HI Titer ≥1:40 at Day 181 | 83.9 [81.48 to 86.17] | 84.0 [81.60 to 86.28]
  B/Victoria HI Titer ≥1:40 at Day 1 | 58.5 [55.42 to 61.57] | 60.4 [57.30 to 63.43]
  B/Victoria HI Titer ≥1:40 at Day 22 | 94.4 [92.79 to 95.72] | 93.3 [91.63 to 94.81]
  B/Victoria HI Titer ≥1:40 at Day 181 | 83.4 [80.90 to 85.66] | 84.3 [81.84 to 86.48]

8. Secondary Outcome: Immunogenicity Endpoint: SCR at Day 22 and Day 181 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains
Description: The SCR defined as the percentage of subjects with either a prevaccination HI titer <1:10 and a postvaccination (Day 22 or Day 181) HI titer ≥1:40, or with either a prevaccination HI titer ≥1:10 and a ≥4-fold increase in postvaccination HI titer.
Time Frame: Day 1 to Day 181
Population: FAS Immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
percentage of participants
  A/H1N1 Day 22 SCR | 80.8 [78.24 to 83.20] | 77.1 [74.34 to 79.65]
  A/H1N1 Day 181 SCR | 64.5 [61.46 to 67.55] | 56.1 [52.94 to 59.24]
  A/H3N2 Day 22 SCR | 63.4 [60.35 to 66.42] | 61.8 [58.65 to 64.79]
  A/H3N2 Day 181 SCR | 39.4 [36.28 to 42.54] | 38.6 [35.51 to 41.72]
  B/Yamagata Day 22 SCR | 42.9 [39.82 to 46.02] | 41.1 [37.99 to 44.19]
  B/Yamagata Day 181 SCR | 22.4 [19.82 to 25.16] | 22.4 [19.86 to 25.19]
  B/Victoria Day 22 SCR | 43.9 [40.86 to 47.08] | 40.6 [37.50 to 43.68]
  B/Victoria Day 181 SCR | 24.3 [21.64 to 27.13] | 23.6 [20.97 to 26.38]

9. Secondary Outcome: Safety Endpoint: Solicited Local and Systemic AEs for 7 Days Following Vaccination
Description: Number and percentage of subjects with solicited local and systemic AEs occurring for 7 days following vaccination
Time Frame: Day 1 through Day 7
Population: Solicited Safety Set, defined as all subjects in the All Exposed Set with any solicited AE data including temperature measurements or use of analgesics/antipyretics
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1020 | 1008
Participants
  Any Solicited AEs | 672 | 541
  Any Solicited Local AEs | 508 | 306
  Any Solicited Systemic AEs | 462 | 403
  Analgesic/Antipyretic Use | 132 | 97

10. Secondary Outcome: Safety Endpoint: All Unsolicited AEs for 21 Days Following Vaccination
Description: The percentage of subjects with at least one unsolicited AE occurring 21 days following vaccination The severity of AEs is based on the maximum severity associated with a Preferred Term for a reported AE. Related AEs include possibly related AEs, probably related AEs and AEs with missing relatedness assessment. The severity and relatedness of AEs were determined by the investigator. For the any AE summary by severity, a subject with multiple AEs is counted according to the highest severity of their reported AEs.
Time Frame: Day 1 through Day 22
Population: Unsolicited Safety Set, defined as all subjects in the All Exposed Set with any unsolicited AE data. Note: Subjects are categorized according to the maximum symptom severity.
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Participants
  Any AE | 169 | 172
  Any AE (Mild) | 116 | 115
  Any AE (Moderate) | 51 | 50
  Any AE (Severe) | 2 | 7
  Related AE | 33 | 32

11. Secondary Outcome: Safety Endpoint: Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Withdrawal From the Study, and Adverse Events of Special Interest (AESIs)
Description: The percentage of subjects with any SAE, AE leading to withdrawal, or AESI during the study period
Time Frame: Day 1 through Day 271
Population: Unsolicited Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Participants
  SAE | 31 | 31
  Related SAE | 0 | 1
  AE leading to study withdrawal | 0 | 1
  AESI | 2 | 0
  Death | 1 | 0

12. Other Pre Specified Outcome: Immunogenicity Endpoint: GMT and GMT Ratio of HI Antibodies at Day 22 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains by Age (Subgroup Analysis)
Description: as for outcome 1
Time Frame: Day 22
Population: FAS Immunogenicity. Subgroup analysis by age (50 to 59 years; 60 to 64 years). Note: Adjusted GMTs are presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Titer
  A/H1N1 (50 to 59 years): number analyzed (Participants) | 609 | 595
  A/H1N1 (50 to 59 years) | 674.25 [622.70 to 730.07] | 565.33 [521.77 to 612.53]
  A/H3N2 (50 to 59 years): number analyzed (Participants) | 609 | 595
  A/H3N2 (50 to 59 years) | 345.83 [317.55 to 376.63] | 319.55 [293.19 to 348.27]
  B/Yamagata (50 to 59 years): number analyzed (Participants) | 609 | 595
  B/Yamagata (50 to 59 years) | 161.27 [150.98 to 172.25] | 149.36 [139.72 to 159.67]
  B/Victoria (50 to 59 years): number analyzed (Participants) | 609 | 595
  B/Victoria (50 to 59 years) | 167.60 [156.68 to 179.27] | 165.81 [154.92 to 177.47]
  A/H1N1 (60 to 64 years): number analyzed (Participants) | 418 | 421
  A/H1N1 (60 to 64 years) | 806.65 [740.51 to 878.70] | 618.90 [567.97 to 674.41]
  A/H3N2 (60 to 64 years): number analyzed (Participants) | 418 | 421
  A/H3N2 (60 to 64 years) | 348.59 [312.82 to 388.45] | 310.23 [278.52 to 345.54]
  B/Yamagata (60 to 64 years): number analyzed (Participants) | 418 | 421
  B/Yamagata (60 to 64 years) | 148.20 [137.62 to 159.59] | 144.34 [134.10 to 155.36]
  B/Victoria (60 to 64 years): number analyzed (Participants) | 418 | 421
  B/Victoria (60 to 64 years) | 119.64 [110.33 to 129.75] | 121.16 [111.79 to 131.32]
Statistical Analysis 1: Comparison: aQIV vs Comparator QIV; A/H1N1 (50 to 59 years); Test type: Other; GMT ratio = 0.838, 95% CI 2-sided [0.751 to 0.936]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; A/H3N2 (50 to 59 years); Test type: Other; GMT ratio = 0.924, 95% CI 2-sided [0.821 to 1.040]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; B/Yamagata (50 to 59 years); Test type: Other; GMT ratio = 0.926, 95% CI 2-sided [0.845 to 1.015]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; B/Victoria (50 to 59 years); Test type: Other; GMT ratio = 0.989, 95% CI 2-sided [0.901 to 1.087]
Statistical Analysis 5: Comparison: aQIV vs Comparator QIV; A/H1N1 (60 to 64 years); Test type: Other; GMT ratio = 0.767, 95% CI 2-sided [0.681 to 0.864]
Statistical Analysis 6: Comparison: aQIV vs Comparator QIV; A/H3N2 (60 to 64 years); Test type: Other; GMT ratio = 0.890, 95% CI 2-sided [0.766 to 1.033]
Statistical Analysis 7: Comparison: aQIV vs Comparator QIV; B/Yamagata (60 to 64 years); Test type: Other; GMT ratio = 0.974, 95% CI 2-sided [0.879 to 1.079]
Statistical Analysis 8: Comparison: aQIV vs Comparator QIV; B/Victoria (60 to 64 years); Test type: Other; GMT ratio = 1.013, 95% CI 2-sided [0.905 to 1.133]

13. Other Pre Specified Outcome: Immunogenicity Endpoint: GMT and GMT Ratio of HI Antibodies at Day 22 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains by Influenza Vaccination History (Subgroup Analysis)
Description: as for outcome 1
Time Frame: Day 22
Population: FAS Immunogenicity. Subgroup analysis by influenza vaccination history (Received at least one influenza vaccination within the previous 3 influenza seasons: yes; no). Note: Adjusted GMTs are presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Titer
  A/H1N1 (yes): number analyzed (Participants) | 586 | 598
  A/H1N1 (yes) | 648.75 [601.45 to 699.78] | 547.54 [508.79 to 589.24]
  A/H3N2 (yes): number analyzed (Participants) | 586 | 598
  A/H3N2 (yes) | 279.61 [257.70 to 303.38] | 282.44 [260.95 to 305.71]
  B/Yamagata (yes): number analyzed (Participants) | 586 | 598
  B/Yamagata (yes) | 116.48 [110.62 to 122.65] | 110.37 [104.98 to 116.04]
  B/Victoria (yes): number analyzed (Participants) | 586 | 598
  B/Victoria (yes) | 101.89 [96.50 to 107.59] | 101.59 [96.39 to 107.07]
  A/H1N1 (no): number analyzed (Participants) | 441 | 418
  A/H1N1 (no) | 755.46 [688.45 to 829.00] | 582.90 [529.83 to 641.28]
  A/H3N2 (no): number analyzed (Participants) | 441 | 418
  A/H3N2 (no) | 389.77 [347.94 to 436.63] | 312.38 [277.97 to 351.06]
  B/Yamagata (no): number analyzed (Participants) | 441 | 418
  B/Yamagata (no) | 188.78 [172.28 to 206.85] | 178.45 [162.38 to 196.12]
  B/Victoria (no): number analyzed (Participants) | 441 | 418
  B/Victoria (no) | 185.31 [168.62 to 203.65] | 186.65 [169.30 to 205.78]
Statistical Analysis 1: Comparison: aQIV vs Comparator QIV; A/H1N1 (yes); Test type: Other; GMT ratio = 0.844, 95% CI 2-sided [0.761 to 0.935]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; A/H3N2 (yes); Test type: Other; GMT ratio = 1.010, 95% CI 2-sided [0.904 to 1.128]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; B/Yamagata (yes); Test type: Other; GMT ratio = 0.948, 95% CI 2-sided [0.883 to 1.016]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; B/Victoria (yes); Test type: Other; GMT ratio = 0.997, 95% CI 2-sided [0.926 to 1.073]
Statistical Analysis 5: Comparison: aQIV vs Comparator QIV; A/H1N1 (no); Test type: Other; GMT ratio = 0.772, 95% CI 2-sided [0.677 to 0.880]
Statistical Analysis 6: Comparison: aQIV vs Comparator QIV; A/H3N2 (no); Test type: Other; GMT ratio = 0.801, 95% CI 2-sided [0.683 to 0.941]
Statistical Analysis 7: Comparison: aQIV vs Comparator QIV; B/Yamagata (no); Test type: Other; GMT ratio = 0.945, 95% CI 2-sided [0.831 to 1.076]
Statistical Analysis 8: Comparison: aQIV vs Comparator QIV; B/Victoria (no); Test type: Other; GMT ratio = 1.007, 95% CI 2-sided [0.881 to 1.151]

14. Other Pre Specified Outcome: Immunogenicity Endpoint: GMT and GMT Ratio of HI Antibodies at Day 22 for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria Vaccine Strains by Comorbidity Risk Score (Subgroup Analysis)
Description: as for outcome 1
Time Frame: Day 22
Population: FAS Immunogenicity. Subgroup analysis by comorbidity risk score (<50; ≥50). Note: Adjusted GMTs are presented.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | aQIV | Comparator QIV
Number analyzed (Participants) | 1027 | 1016
Titer
  A/H1N1 (Comorbidity Risk Score <50): number analyzed (Participants) | 912 | 918
  A/H1N1 (Comorbidity Risk Score <50) | 715.26 [671.75 to 761.60] | 586.42 [550.95 to 624.16]
  A/H3N2 (Comorbidity Risk Score <50): number analyzed (Participants) | 912 | 918
  A/H3N2 (Comorbidity Risk Score <50) | 337.43 [314.06 to 362.53] | 314.75 [293.14 to 337.96]
  B/Yamagata (Comorbidity Risk Score <50): number analyzed (Participants) | 912 | 918
  B/Yamagata (Comorbidity Risk Score <50) | 150.17 [142.37 to 158.40] | 145.98 [138.44 to 153.93]
  B/Victoria (Comorbidity Risk Score <50): number analyzed (Participants) | 912 | 918
  B/Victoria (Comorbidity Risk Score <50) | 139.76 [132.15 to 147.82] | 141.58 [133.93 to 149.68]
  A/H1N1 (Comorbidity Risk Score ≥50): number analyzed (Participants) | 115 | 98
  A/H1N1 (Comorbidity Risk Score ≥50) | 812.59 [681.59 to 968.76] | 573.86 [473.11 to 696.06]
  A/H3N2 (Comorbidity Risk Score ≥50): number analyzed (Participants) | 115 | 98
  A/H3N2 (Comorbidity Risk Score ≥50) | 453.60 [368.59 to 558.20] | 333.16 [265.15 to 418.62]
  B/Yamagata (Comorbidity Risk Score ≥50): number analyzed (Participants) | 115 | 98
  B/Yamagata (Comorbidity Risk Score ≥50) | 198.10 [172.89 to 227.00] | 153.05 [131.91 to 177.58]
  B/Victoria (Comorbidity Risk Score ≥50): number analyzed (Participants) | 115 | 98
  B/Victoria (Comorbidity Risk Score ≥50) | 174.79 [151.43 to 201.74] | 158.12 [135.26 to 184.85]
Statistical Analysis 1: Comparison: aQIV; A/H1N1 (Comorbidity Risk Score <50); Test type: Other; GMT ratio = 0.820, 95% CI 2-sided [0.752 to 0.894]
Statistical Analysis 2: Comparison: aQIV vs Comparator QIV; A/H3N2 (Comorbidity Risk Score <50); Test type: Other; GMT ratio = 0.933, 95% CI 2-sided [0.846 to 1.029]
Statistical Analysis 3: Comparison: aQIV vs Comparator QIV; B/Yamagata (Comorbidity Risk Score <50); Test type: Other; GMTratio = 0.972, 95% CI 2-sided [0.904 to 1.046]
Statistical Analysis 4: Comparison: aQIV vs Comparator QIV; B/Victoria (Comorbidity Risk Score <50); Test type: Other; GMT ratio = 1.013, 95% CI 2-sided [0.938 to 1.094]
Statistical Analysis 5: Comparison: aQIV vs Comparator QIV; A/H1N1 (Comorbidity Risk Score ≥50); Test type: Other; GMT ratio = 0.706, 95% CI 2-sided [0.553 to 0.902]
Statistical Analysis 6: Comparison: aQIV vs Comparator QIV; A/H3N2 (Comorbidity Risk Score ≥50); Test type: Other; GMT ratio = 0.734, 95% CI 2-sided [0.549 to 0.982]
Statistical Analysis 7: Comparison: aQIV vs Comparator QIV; B/Yamagata (Comorbidity Risk Score ≥50); Test type: Other; GMT ratio = 0.773, 95% CI 2-sided [0.638 to 0.935]
Statistical Analysis 8: Comparison: aQIV vs Comparator QIV; B/Victoria (Comorbidity Risk Score ≥50); Test type: Other; GMT ratio = 0.905, 95% CI 2-sided [0.739 to 1.107]

ADVERSE EVENTS:
Time Frame: SAEs: Day 1 through Day 271; nonserious unsolicited AEs: Day 1 through Day 22; solicited AEs: Day 1 through Day 7
Description: Number and percentage of subjects with SAEs and other AEs (ie, nonserious unsolicited AEs and solicited AEs)
  All-cause mortality and SAEs are reported for the Unsolicited Safety Set. In the category of "Other Adverse Events", no nonserious unsolicited AEs were reported at a frequency >5%; therefore, only solicited AEs occurring at a frequency >5% in the Solicited Safety Set are reported in this section.
Arm/Group | aQIV | Comparator QIV
All-Cause Mortality (participants affected / at risk) | 1/1027 | 0/1016
Serious Adverse Events (participants affected / at risk) | 31/1027 | 31/1016
Other Adverse Events (participants affected / at risk) | 660/1020 | 519/1008
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (N=1027) | Comparator QIV (N=1016)
COVID-19 (Infections and infestations) | 3 | 0
Abscess limb (Infections and infestations) | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Huerthle cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Bladder injury (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Hernia pain (General disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Middle ear adhesions (Ear and labyrinth disorders) | 0 | 1
Allergy to metals (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (N=1020) | Comparator QIV (N=1008)
Diarrhea (Gastrointestinal disorders) | 81 | 71
Nausea (Gastrointestinal disorders) | 74 | 44
Chills (General disorders) | 67 | 55
Fatigue (General disorders) | 301 | 245
Induration (General disorders) | 81 | 35
Injection site pain (General disorders) | 480 | 283
Decreased appetite (Metabolism and nutrition disorders) | 62 | 48
Arthralgia (Musculoskeletal and connective tissue disorders) | 140 | 95
Myalgia (Musculoskeletal and connective tissue disorders) | 133 | 73
Headache (Nervous system disorders) | 226 | 206
Erythema (Skin and subcutaneous tissue disorders) | 80 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Seqirus will generally support publication of multicenter studies only in their entirety and not as individual center data.

Seqirus must be notified of any intent to publish data collected from the study and prior approval from Seqirus must be obtained prior to submission for publication.

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT05044195/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT05044195/SAP_001.pdf